CLINICAL TRIAL: NCT05671315
Title: A Prospective, Randomized, Open-label, Multicenter Study to Evaluate the Peginterferon, Comparing to Nucleos(t)Ide Analogues, in Reducing the Incidence of HCC in Chronic Hepatitis B Patients With Intermediate to High Liver Cancer Risks
Brief Title: A Prospective Study to Evaluate Peginterferon in Reducing the Incidence of HCC in CHB Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qing XIe (Other)
Responsible Party: Sponsor-Investigator, Qing XIe, Director of Department of Infectious Disease, Rui Jin Hospital, Ruijin Hospital
Organization: Ruijin Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Paradise
Record Dates: First submitted 2020-03-15; First posted 2023-01-04 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Chronic Hepatitis B; Intermediate to High Risk of HCC
Keywords: Chronic Hepatitis B; Hepatocellular Carcinoma; Peginterferon; Nucleos(t)ide analogue
MeSH Terms: conditions — Hepatitis B, Chronic; Carcinoma, Hepatocellular | interventions — peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined treatment group (Experimental): Peginterferon alfa-2b Injection combined Nucleos (t) ide Analogue therapy
  Interventions: Drug: Peginterferon alfa-2b Injection, Nucleos (t) ide Analogue
- Monotherapy group (Active Comparator): Nucleos (t) ide Analogue monotherapy
  Interventions: Drug: Nucleos(t)ide analogue

INTERVENTIONS:
Drug: Peginterferon alfa-2b Injection, Nucleos (t) ide Analogue — 1.Peginterferon alfa-2b injection: 180μg, subcutaneously inject, once a week, from week 1 to Week 48.
  2, NAs: Dose please follow the approved dosage, once daily, from the first day until when discontinuation is indicated.
  NAs Discontinuation Criteria: A total course of treatment is recommended for at least 4 years, and discontinuation may be considered if HBV DNA is below the lower limit of detection, Alanine aminotransferase renormalization, and HBeAg serological conversion, and remain unchanged (test every 6 months) during a consolidation therapy for at least 3 years. However, a prolonged course of treatment may reduce relapse.
  Arms: Combined treatment group
Drug: Nucleos(t)ide analogue — NAs: Dose please follow the approved dosage, once daily, from the first day until when discontinuation is indicated.
  NAs Discontinuation Criteria: A total course of treatment is recommended for at least 4 years, and discontinuation may be considered if HBV DNA is below the lower limit of detection, Alanine aminotransferase renormalization, and HBeAg serological conversion, and remain unchanged (test every 6 months) during a consolidation therapy for at least 3 years. However, a prolonged course of treatment may reduce relapse.
  Arms: Monotherapy group

SUMMARY:
China's new cases and deaths of hepatocellular carcinoma (HCC) rank first in the world. hepatocellular carcinoma is the third most morbid, second-most mortal malignancy in China. Up to 80% of hepatocellular carcinoma patients caused by HBV infection. Antiviral therapy can significantly reduce the incidence and mortality of hepatocellular carcinoma in patients with chronic hepatitis B (CHB), hinder the progression of liver disease, and effectively control the disease. However, studies in recent years have found that long-term therapy with Nucleos(t)ide analogue (NAs) cannot completely eliminate the risk of liver cancer in patients with chronic hepatitis B. In addition, a number of retrospective studies at home and abroad have shown that compared with long-term oral NAs, peginterferon can significantly reduce the risk of hepatocellular carcinoma in patients with chronic hepatitis B. However, there is limit prospective studies.

This multicenter, randomized, open-label, controlled trial study is aim to evaluate the pegylated interferon alfa-2b injection in comparing to NAs in reducing the incidence of hepatocellular carcinoma, to provide evidences for new management and treatment strategy options for improving clinical outcomes for the chronic hepatitis B patients. About 267 chronic hepatitis patients with intermediate to high risk of liver cancer who are now receiving nucleoside therapy will be enrolled. Subjects will be randomized into the peginterferon combined NAs group and the NAs monotherapy group at a ratio of 2:1. Level of HBsAg, proportion of patients with HBsAg clearance and seroconversion, incidence of liver cirrhosis and hepatocellular carcinoma will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 60 years and no gender limit (including 18 and 60 years).
* HBsAg positive for more than 6 months.
* Patients with intermediate to high liver cancer risks. Refers to if at least one of the following items is met.

  * Male patient aged above 40 years.
  * Patients with a history of cirrhosis and/or family history of liver cancer.
  * Patients with metabolic diseases, such as diabetes, fatty liver, etc.
  * Any liver cancer assessment model of chronic hepatitis B patients suggested that liver cancer was at intermediate to high risk.
* Have received Nucleos(t)ide analogue treatment for more than 24 weeks, and currently receiving Nucleos(t)ide analogue, while HBV DNA is undetectable (HBV DNA below 300 IU/mL or 1000 copies/mL).
* Urine and/or serum pregnancy test within 24 hours prior to the first dose must be negative for female patients of childbearing potential.
* Understand and voluntarily sign informed consent form.

Exclusion Criteria:

* Patients co-infected with active hepatitis A, hepatitis C, hepatitis D, hepatitis E or HIV.
* Patients who have previously received interferon therapy.
* Alpha-fetoprotein greater than 100 ng/mL at screening, or liver imaging suggestive of liver tumor.
* Decompensated liver disease (Child-Pugh score ≥ 5).
* Pregnant or lactating women or patients planning to become pregnant or cannot to take contraception during the study.
* Neutrophil count < 1.5 x 109/L, platelet count < 90 x 109 cells/L, or Creatinine 1.5 times higher than the upper limit of normal.
* Patients with severe psychiatric history, particularly depression.
* History of immune-mediated disease or levels of autoimmune antibodies markedly elevated.
* Patients with severe diseases in major organ, such as heart, lung, kidney, brain, blood, etc., and patients with malignancies.
* Patients with poorly controlled diabetes, hypertension, and thyroid disease.
* Patients with history of severe retinopathy or other evidence of retinopathy.
* Patient who ever received organ transplantation, or planning to receive organ transplantation.
* Patients who are allergic to interferon or any of its ingredients.
* Other circumstances that the investigator deems inappropriate to participate in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 267 (Estimated)
Dates: Start 2019-07-03 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change of HBsAg level compared to baseline | week 48 of treatment

SECONDARY OUTCOMES:
Proportion of patients with HBsAg clearance | At week 48 of treatment and 5 years of follow up
Proportion of patients with HBsAg seroconversion | At week 48 of treatment and 5 years of follow up
Proportion of patients with change of liver stiffness measurement (LSM) | At week 48 of treatment and 5 years of follow up
Incidence of liver cirrhosis and hepatocellular carcinoma | At week 48 of treatment and 5 years of follow up

CONTACTS AND LOCATIONS:
Overall Officials: Qing Xie, Principal Investigator — Ruijin Hospital, Shanghai
Locations (9):
- China (9):
  - The Public Health Clinical Center Of Chengdu, Chengdu
  - The First Affiliated Hospital of USTC Anhui Provincial Hospital, Hefei
  - The Affiliated Hospital of Qingdao University, Qingdao
  - Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shanghai Ninth People's Hospital Shanghai Jiao Tong University School of Medicine, Shanghai
  - Tongren Hospital Shanghai Jiao Tong University School of Medicine, Shanghai
  - The Fifth People's Hospital Of Suzhou, Suzhou
  - Xiamen Hospital of Traditional Chinese Medicin, Xiamen
  - The Tirth Affiliated Hospital Of Xinxiang Medical University, Xinxiang

REFERENCES:
- [Derived] Jiang S, Guo S, Huang Y, Xu J, Li Y, Zeng Y, Guo Y, Ouyang L, Zhu C, Zhao W, Zhang Q, Guo Q, Xin H, Xie Q. Interim analysis of the PARADISE study: Benefits of add-on peginterferon-alpha in NA-treated patients with CHB. Antiviral Res. 2024 Jun;226:105892. doi: 10.1016/j.antiviral.2024.105892. Epub 2024 Apr 23. PMID 38663455